CLINICAL TRIAL: NCT02477631
Title: The Effect of Treatment With the Oral Iron Chelator Deferiprone on the Oxidative Stress of Blood Cells and on Iron Overload Status in Transfusion Dependent, Iron-overloaded Patients With Low Risk Myelodysplastic Syndrome
Brief Title: Effect of Deferiprone on Oxidative-Stress and Iron-Overload in Low Risk Transfusion-Dependent MDS Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Hadassah Medical Organization (Other); Tel Aviv Medical Center (Other); Kaplan Medical Center (Other); Ziv Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Drorit Merkel, Senior physician in the Hematology wing, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-15-1908-DM-CTIL
Record Dates: First submitted 2015-05-11; First posted 2015-06-23 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Myelodysplastic Syndrome With Low-grade Lesions; Iron Overload Due to Repeated Red Blood Cell Transfusions
Keywords: Myelodysplastic syndrome; oxidative stress; labile plasma iron
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Deferiprone; Long Interspersed Nucleotide Elements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deferiprone (Experimental): patient treated with study drug
  Interventions: Drug: Deferiprone

INTERVENTIONS:
Drug: Deferiprone — This is a single-arm, open-label, multi-center study in 20 patients with MDS. All participants will be treated with deferiprone for up to 4 months.
  Other Names: L1, Ferriprox

SUMMARY:
The effect oral iron chelator Deferiprone on the Oxidative stress and on Iron Overload status in transfusion dependent, iron-overloaded low risk MDS patients;

Primary Objective:

• To evaluate the effect of Deferiprone on oxidative stress parameter - Reactive oxygen species (ROS).

Secondary Objectives:

* To evaluate the effect of Deferiprone on other oxidative stress parameters

  1. Reduced glutathione
  2. Membrane lipid peroxidation
  3. External phosphatidylserine
* To evaluate the change from baseline to last visit in parameters of iron load.

  1. Serum ferritin (despite ongoing RBC transfusions during the study period).
  2. LIP
  3. LPI
  4. serum hepcidin
* To evaluate the change from one month preceding baseline visit to last month on study in transfusion requirements.
* To monitor safety measures:

  1. Adverse events (AEs).
  2. Number of discontinuations due to AEs

Study design:

Single-arm, open-label, multi-center study in 20 iron-overloaded patients with low risk MDS. All participants will be treated with deferiprone for up to 4 months. Patients will have complete blood count monitored weekly, and will visit the site monthly for assessments of safety and efficacy.

DETAILED DESCRIPTION:
INTRODUCTION 1.1 Background Myelodysplastic syndrome (MDS) is characterized by deficiencies in blood cell production that can lead to anemia, which may necessitate regular transfusions of red blood cells (RBCs) as supportive therapy. While this treatment can be life-saving, since the body has no natural means of removing the excess iron introduced through the intake of RBCs, a consequence can be accumulation of excess iron, including labile iron, in the plasma (as labile plasma iron, LPI, the pathological form of non-transferrin-bound iron) and in cells. The cellular labile iron pool (LIP) is known to participate in biochemical reactions that generate free oxygen radicals, resulting in oxidative stress and cell and tissue damage. A certain percentage of patients with MDS develop signs and symptoms resulting from iron overload، and oxidative stress markers have been observed in the blood cells of such patients. Progressive iron overload can lead to organ toxicity and cardiac disease. Reduction of LIP would reduce the generation of tissue-damaging free oxygen radicals and thereby help prevent morbidity and mortality; however, iron chelation therapy has not been part of the standard of care for this population. It should be noted that While the LPI level provide a momentarily "snapshot" of the iron status and it rapidly changes due to nutrition, transfusion or chelation, the LIP represent long-term accumulation. Both parameters complement each other in analogy to hemoglobin A1C and glucose measurements in patients with Diabetes mellitus).

There has been some exploration of the use of the oral iron chelators deferasirox and deferiprone in MDS patients , with indications of efficacy as assessed by iron reduction, decreased need for transfusions, or increased survival. However, it is difficult to draw clear conclusions from the literature as there was high variability in these investigations, not only in type of chelator but in study design, severity of disease, and endpoints studied. The safety profiles reported in the literature for MDS patients are similar to those seen in thalassemia patients. However, for patients at later stages of the disease who are at high risk of death from AML or other causes within 5 years, the benefit of chelation may be minimal. What emerges from the literature is that because of the progression of the disease, iron chelation is likelier to be of more benefit to patients with a less severe form of MDS who have an expectation of 5 years or more of survival but who also have the likelihood of long-term RBC transfusion dependency, with the accompanying risk of iron overload.

1.2 Deferiprone Deferiprone (active ingredient 3-hydroxy-1,2-dimethylpyridin-4-one) is a bidentate iron chelator that preferentially binds trivalent iron (Fe3+) in a 3:1 (deferiprone : iron) complex. Its effectiveness in the treatment of patients with iron overload has been assessed by urinary iron excretion, sequential measurements of serum ferritin levels, iron concentration in the liver and in the heart, and clinical outcomes such as the ability to prevent iron-induced cardiac disease and prolong survival in transfused patients with thalassemia.

1.2.1 Side effects of Deferiprone The safety profile of deferiprone in patients with thalassemia has been extensively characterized in clinical trials. Based on the Summary of Product Characteristics,apart from chromaturia, which is due to iron excretion and is harmless, the most commonly reported adverse events seen in clinical trials have been nausea, vomiting, abdominal pain, increased alanine aminotransferase, arthralgia, and neutropenia, defined as a confirmed absolute neutrophil count (ANC) less than 1.5×109/L. The most significant serious adverse event (SAE) associated with deferiprone use is severe neutropenia, also known as agranulocytosis, which is defined as a confirmed ANC less than 0.5×109/L.

In a clinical trial in which 19 multi-transfused MDS patients were treated with the oral iron chelator deferasirox for 3 months, a significant decrease in free iron species was observed in the plasma and cells, which was associated with amelioration of the parameters of oxidative stress. Another finding was a gradual increase in the levels of the iron regulatory hormone hepcidin, which could also reflect amelioration of oxidative stress. However, many MDS patients, particularly older ones, are unable to tolerate treatment with deferasirox, mainly due to renal and/or gastrointestinal side effects. The proposed clinical trial is a similar study that will look at the safety and efficacy of deferiprone in iron overloaded, blood dependent MDS patients.

2 STUDY DESIGN This is a single-arm, open-label, multi-center study in 20 patients with MDS. All participants will be treated with deferiprone for up to 4 months. Patients will have blood counts monitored weekly, and will visit the site monthly for assessments of safety and efficacy. The schedule of study procedures is shown and details are provided in Section 5.1.

The daily dosage of deferiprone for each patient will be up to a maximum dose of 100 mg/kg, divided into 3 equal doses (t.i.d.) of 33.3 mg/kg. To minimize the gastrointestinal side effects that some deferiprone recipients experience when starting treatment, the initial dosage will be a total of 50 mg/kg/day (16.7 mg/kg t.i.d. For patients responding to treatment, there will be an option to continue the study drug for one more year.

3 STUDY POPULATION 3.1 Number of Patients A total of 20 MDS patients 3.2 Treatment Interruptions Patients should be advised to immediately report any symptoms indicative of infection such as fever, sore throat, or flu-like symptoms. If a patient develops neutropenia, fever, or any type of infection, Deferiprone must be interrupted immediately and neutrophil count should be obtained and monitored more frequently.

3.3 Concomitant medications In general, concomitant medications and therapies deemed necessary for the supportive care and safety of the patient are allowed. The administration of any anticancer agents including chemotherapy and biologic agents is permitted. The use of other concurrent iron chelating agents or iron supplements or investigational drugs is not allowed. The use of blood products transfusions or erythroid growth factor is permitted at investigator's discretion.

3.4 Study treatment discontinuation

The following events will be considered as reasons for discontinuation:

* Intolerable adverse effects that are judged by the investigator to be detrimental to the patient.
* Participation in another investigational drug trial
* Loss to follow up
* Patient withdrawal of consent 4 STUDY TREATMENTS Deferiprone is provided as 500 mg film-coated scored tablets, taken orally 3 times a day. It can also be provided as an oral solution of deferiprone 100mg/ml. The drug can be taken with or without food, as per the investigator's recommendation.

  5 MEASUREMENTS AND EVALUATIONS 5.1 Efficacy Measurements

Primary Objective:

• To evaluate the effect of Deferiprone on oxidative stress parameter - Reactive oxygen species (ROS).

Secondary Objectives:

* To evaluate the effect of Deferiprone on other oxidative stress parameters

  1. Reduced glutathione
  2. Membrane lipid peroxidation
  3. External phosphatidylserine
* To evaluate the change from baseline to last visit in parameters of iron load.

  1. Serum ferritin (despite ongoing RBC transfusions during the study period).
  2. LIP
  3. LPI
  4. serum hepcidin
* To evaluate the change from one month preceding baseline visit to last month on study in transfusion requirements.
* To monitor safety measures:

  1. Adverse events (AEs).
  2. Number of discontinuations due to AEs

5.1.1 Oxidative stress parameters Blood samples for the assessment of oxidative stress parameters will be collected at baseline and at each monthly visit. Samples will be taken at similar times for all patients, prior to first morning dose of Deferiprone. Blood samples will be collected into 2 test tubes, 2cc in each tube. One test tube with heparin and sent in the same day or the day after in a temperature of 40c to the laboratory of Prof. Fibach.

Oxidative status (as well as LIP) will be analyzed using flow cytometry techniques. Red blood cells (RBCs) and platelets will be analyzed for all tests of oxidative stress, while polymorphonuclear leucocytes will be analyzed only for ROS and Iron Overload Iron overload will be evaluated by measuring serum ferritin, LIP, LPI, and serum hepcidin.

Blood samples for serum ferritin will be collected at baseline, and each monthly visit, and end of study.

Blood samples for the assessment of LIP, LPI will be collected at baseline and each monthly visit, and will be sent to Hadassah University Hospital, Jerusalem (LIP) and to Aferrix Ltd., Rehovot (LPI), Israel for analysis.

Two-ml blood samples will be drawn in heparin for the assessment of oxidative stress parameters, LIP and LPI. For serum hepcidin, 2-ml samples will be drawn without an anti-coagulant. All samples will be kept and transported on ice, on the same day, to Hadassah hospital, Ein-Kerem, Jerusalem. Upon arrival to Hadassah, cells, plasma and serum, as required, will be separated. Cellular measurements will be performed on the day of arrival or the next day. The plasma and serum will be kept frozen until assayed for LPI and serum ferritin, respectively.

Serum samples for the assessment of hepcidin levels will be collected at baseline and each monthly visit. All samples will be sent to the laboratory of Dr. Domenico Girelli in Verona, Italy, for analysis after being kept until the end of the study in prof' Fibach laboratory.

5.1.2 Transfusion Requirements At each visit, patients will be queried about the receipt of RBC transfusions from last visit: type of transfusion, the volume (number of transfusions) of blood received. Details will be obtained from the site's blood bank.

. 5.1.3 Laboratory Measurements

Samples for the following laboratory safety assessments will be taken a designated time points throughout the study:

* Hematology (weekly): hemoglobin, WBC count, ANC, and platelet count
* Biochemistry (screening, baseline, and each monthly visit): total protein, GGT, lactate dehydrogenase (LDH), sodium, potassium, chloride, glucose, total and direct bilirubin, AST, ALT, albumin, blood urea nitrogen, calcium, creatinine, uric acid, alkaline phosphatase, and amylase
* Serum pregnancy test: screening, baseline, and each monthly visit

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 years
2. Have a documented diagnosis of MDS according to WHO 2008 classification (see appendix I), with an International Prognostic Scoring System (IPSS-R) (see Appendix II) of very low, low or intermediate risk.
3. Life expectancy of at least 1 year
4. Serum ferritin level > 1000 ng/mL
5. Prior receipt of ≥20 RBC units
6. Females of childbearing potential must have a negative pregnancy test result month prior to start of dosing, In addition, if applicable, they must:

   * Use an effective method of contraception according to local requirements, during the study and within 30 days following their last dose of study medication, OR
   * Have had a tubal ligation (supporting evidence required), OR
   * Have had a hysterectomy (supporting evidence required), OR
   * Participate in a non-heterosexual lifestyle, OR
   * Have a male sexual partner who has been sterilized (supporting evidence required)
7. Non-sterilized heterosexual males and/or their partners must agree to use an effective method of contraception during the study and for 30 days following their last dose of study medication
8. All patients and/or their authorized legal representatives must provide signed and dated written informed consent prior to the first study intervention, and patients must be able to adhere to study restrictions, appointments, and evaluation schedules

Exclusion Criteria:

1. IPSS-R prognosis of high and very high risk (to avoid the confounding influence of a high blast count)
2. Unable or unwilling to undergo a 7-day washout period if currently being treated with deferoxamine or deferasirox
3. Evidence of abnormal liver function (serum ALT level > 5 times upper limit of normal or creatinine level >2 times upper limit of normal)
4. A serious, unstable illness, as judged by the investigator, during the past 3 months before screening, including but not limited to: hepatic, renal, gastro-enterologic, respiratory, cardiovascular, endocrinologic, neurologic, or immunologic disease
5. Myocardial infarction, cardiac arrest, or cardiac failure within 1 year before screening
6. QT interval prolongation on ECG
7. Occurrences of severe neutropenia/agranulocytosis (absolute neutrophil count < 0.5 x 109/L
8. History of allergy or sensitivity to deferiprone or related compounds or to other components of the formulation
9. Receipt of any investigational products within the past 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication
10. Participation in any investigational clinical study, other than observational, within the past 30 days; or plans to participate in such a study at any time from the day of enrollment until 30 days post-treatment in the current study
11. History of drug or alcohol abuse within the last 6 months
12. Presence of any medical, psychological, or psychiatric condition which in the opinion of the investigator would cause participation in the study to be unwise
13. Pregnant, breastfeeding, or planning to become pregnant during the study period.
14. Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication
15. Identified as an investigator or other site staff directly affiliated with this study, or an immediate family member (spouse, parent, child, or sibling, whether biological or legally adopted) of either of the above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of deferiprone on oxidative stress parameter ROS in iron overloaded and blood dependent patients with MDS. | 4 months
  The change from baseline to end of study in ROS

SECONDARY OUTCOMES:
To evaluate the effect of Deferiprone on other oxidative stress parameters-Reduced glutathione | 4 months
  The change from baseline to end of study in Reduced glutathione
To evaluate the effect of Deferiprone on other oxidative stress-Membrane lipid peroxidation | 4 months
  The change from baseline to end of study in lipid peroxidation
To evaluate the effect of Deferiprone on other oxidative stress parameters - External phosphatidylserine | 4 months
  The change from baseline to end of study in External phosphatidylserine
To evaluate the change from baseline to last visit in parameters of iron load-serum ferritin levels (despite ongoing RBC transfusions during the study period). | 4 months
  The change from baseline to end of study in serum ferritin levels
To evaluate the change from baseline to last visit in parameters of iron load- LIP | 4 months
  The change from baseline to end of study in serum LIP levels
To evaluate the change from baseline to last visit in parameters of iron load- LPI | 4 months
  The change from baseline to end of study in serum LPI levels
To evaluate the change from baseline to last visit in parameters of iron load- serum hepcidin | 4 months
  The change from baseline to end of study in serum hepcidin levels
To evaluate the change from one month preceding baseline visit to last month on study in transfusion requirements. | 4 months

OTHER OUTCOMES:
Adverse events (AEs) | 4 months
  Frequency, severity, time to onset, duration, and relatedness to study product and number of discontinuations due to AEs

CONTACTS AND LOCATIONS:
Overall Officials: Drorit Merkel, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Chim Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Greenberg PL, Young NS, Gattermann N. Myelodysplastic syndromes. Hematology Am Soc Hematol Educ Program. 2002:136-61. doi: 10.1182/asheducation-2002.1.136. PMID 12446422
- [Background] Hellstrom-Lindberg E. Management of anemia associated with myelodysplastic syndrome. Semin Hematol. 2005 Apr;42(2 Suppl 1):S10-3. doi: 10.1053/j.seminhematol.2005.01.002. No abstract available. PMID 15846579
- [Background] Hershko C, Link G, Cabantchik I. Pathophysiology of iron overload. Ann N Y Acad Sci. 1998 Jun 30;850:191-201. doi: 10.1111/j.1749-6632.1998.tb10475.x. PMID 9668540
- [Background] Farquhar MJ, Bowen DT. Oxidative stress and the myelodysplastic syndromes. Int J Hematol. 2003 May;77(4):342-50. doi: 10.1007/BF02982641. PMID 12774921
- [Background] Choi SO, Cho YS, Kim HL, Park JW. ROS mediate the hypoxic repression of the hepcidin gene by inhibiting C/EBPalpha and STAT-3. Biochem Biophys Res Commun. 2007 Apr 27;356(1):312-7. doi: 10.1016/j.bbrc.2007.02.137. Epub 2007 Mar 5. PMID 17349976
- [Result] Gattermann N, Rachmilewitz EA. Iron overload in MDS-pathophysiology, diagnosis, and complications. Ann Hematol. 2011 Jan;90(1):1-10. doi: 10.1007/s00277-010-1091-1. Epub 2010 Oct 12. PMID 20938663
- [Result] Ghoti H, Amer J, Winder A, Rachmilewitz E, Fibach E. Oxidative stress in red blood cells, platelets and polymorphonuclear leukocytes from patients with myelodysplastic syndrome. Eur J Haematol. 2007 Dec;79(6):463-7. doi: 10.1111/j.1600-0609.2007.00972.x. Epub 2007 Nov 1. PMID 17976187
- [Result] Smeets ME, Vreugdenhil G, Holdrinet RS. Improvement of erythropoiesis during treatment with deferiprone in a patient with myelofibrosis and transfusional hemosiderosis. Am J Hematol. 1996 Mar;51(3):243-4. doi: 10.1002/(SICI)1096-8652(199603)51:33.0.CO;2-H. No abstract available. PMID 8619408
- [Result] Cermak J. Erythropoietin administration may potentiate mobilization of storage iron in patients on oral iron chelation therapy. Hemoglobin. 2006;30(1):105-12. doi: 10.1080/03630260500455375. PMID 16540422
- [Result] Payne KA, Rofail D, Baladi JF, Viala M, Abetz L, Desrosiers MP, Lordan N, Ishak K, Proskorovsky I. Iron chelation therapy: clinical effectiveness, economic burden and quality of life in patients with iron overload. Adv Ther. 2008 Aug;25(8):725-42. doi: 10.1007/s12325-008-0085-z. PMID 18704280
- [Result] Cermak J, Jonasova A, Vondrakova J, Walterova L, Hochova I, Siskova M, Neuwirtova R. Efficacy and safety of administration of oral iron chelator deferiprone in patients with early myelodysplastic syndrome. Hemoglobin. 2011;35(3):217-27. doi: 10.3109/03630269.2011.578515. PMID 21599434
- [Result] Cermak J, Jonasova A, Vondrakova J, Cervinek L, Belohlavkova P, Neuwirtova R. A comparative study of deferasirox and deferiprone in the treatment of iron overload in patients with myelodysplastic syndromes. Leuk Res. 2013 Dec;37(12):1612-5. doi: 10.1016/j.leukres.2013.07.021. Epub 2013 Aug 9. PMID 23937987
- [Result] Kersten MJ, Lange R, Smeets ME, Vreugdenhil G, Roozendaal KJ, Lameijer W, Goudsmit R. Long-term treatment of transfusional iron overload with the oral iron chelator deferiprone (L1): a Dutch multicenter trial. Ann Hematol. 1996 Nov;73(5):247-52. doi: 10.1007/s002770050236. PMID 8959943
- [Result] Telfer PT, Prestcott E, Holden S, Walker M, Hoffbrand AV, Wonke B. Hepatic iron concentration combined with long-term monitoring of serum ferritin to predict complications of iron overload in thalassaemia major. Br J Haematol. 2000 Sep;110(4):971-7. doi: 10.1046/j.1365-2141.2000.02298.x. PMID 11054091
- [Result] Olivieri NF, Nathan DG, MacMillan JH, Wayne AS, Liu PP, McGee A, Martin M, Koren G, Cohen AR. Survival in medically treated patients with homozygous beta-thalassemia. N Engl J Med. 1994 Sep 1;331(9):574-8. doi: 10.1056/NEJM199409013310903. PMID 8047081